CLINICAL TRIAL: NCT04086524
Title: A Patch Free Treatment for Young Children With Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Retina Foundation of the Southwest (Other); McGill University (Other); Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Ben Thompson, Professor, University of Waterloo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12345; 3600-105 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Amblyopia; Binocular Vision Disorder
Keywords: Amblyopia; Binocular treatment; Visual acuity; Stereopsis; Motor function
MeSH Terms: conditions — Amblyopia | interventions — Working Conditions

STUDY DESIGN:
Intervention Model Description: TREATMENT = 2 weeks of treatment (additional 2 weeks if they agree) CONTROL = 2 weeks patching, 2 weeks treatment
Who Masked: Outcomes Assessor
Masking Description: Study team members measuring outcome variables will be masked to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Binocular cartoon treatment at home (Experimental): Participants will view a dichoptic binocular cartoon (provided by BBC) on the Nintendo 3DS-XL at home. They will continue to watch the cartoon for 60 minutes, 4 times a week, for 2 weeks. After 2 weeks, they will be given the option to continue for an additional 2 weeks (total of 4 weeks). Watching the cartoon does not require any special glasses. They will discontinue patching during this time.
  Interventions: Other: Binocular cartoon treatment at home
- Control group (Active Comparator): Participants will patch for 2 hours every day at home. After 2 weeks, they will be given the option to crossover to the teratment group for an additional 2 weeks (total of 4 weeks). Patching is a common treatment for amblyopia, often considered the "golden standard." It is the most common comparison as a "control" group in amblyopia and vision therapy literature.
  Interventions: Other: Patching
- Binocular cartoon treatment in office (Experimental): Participants will view a dichoptic binocular cartoon (provided by BBC) on the Nintendo 3DS-XL in office. They will continue to watch the cartoon for 60 minutes, 4 times a week, for 2 weeks. After 2 weeks, they will be given the option to continue for an additional 2 weeks (total of 4 weeks). Watching the cartoon does not require any special glasses. They will discontinue patching during this time.
  Interventions: Other: Binocular cartoon treatment in office

INTERVENTIONS:
Other: Binocular cartoon treatment at home — see arm description.
  Arms: Binocular cartoon treatment at home
Other: Patching — see arm description
  Other Names: occlusion therapy; penalization
  Arms: Control group
Other: Binocular cartoon treatment in office — see arm description.
  Arms: Binocular cartoon treatment in office

SUMMARY:
The purpose of this study is to test whether a binocular treatment can improve vision and motor function in young children with amblyopia. The proposed treatment is an animation series that has been modified so that different characters in the animation are presented to each eye. The contrast of the images shown to the amblyopic eye is higher than the contrast of the images shown to the fellow eye. The aim of the treatment is to promote co-operation between the two eyes and improve visual and motor outcomes. We will compare the benefits of this binocular treatment to patching, whereby the better eye is occluded with an eye patch for two hours per day to force the usage of the weaker eye. We hypothesize that the binocular treatment will improve vision and motor outcomes in young children with amblyopia, and that these improvements will be superior to any effects of patching.

DETAILED DESCRIPTION:
This is a prospective study with study sites in Ontario, Canada (University of Waterloo); Quebec, Canada (University of McGill); Texas, United States of America (Retina Foundation of the Southwest); and Queensland, Australia (Queensland University of Technology). There are three study conditions. 1) binocular treatment at home, 2) binocular treatment in office and, 3) standard patching therapy.

Participants will be recruited from university-affiliated clinics and local clinical practices. Following full informed consent, participants will complete baseline testing to confirm eligibility and provide pre-treatment measurements of visual acuity, stereopsis, interocular suppression and motor function. Eligible participants will then be randomized to either binocular treatment or patching.

The treatment consists of dichoptically presented children's animations with all characters seen by the amblyopic eye and only a subset of characters seen by the fellow eye. Images shown to the amblyopic eye will be presented at 100% contrast and images presented to the fellow eye will be presented at 20% contrast on session 1 and contrast will increment by 10% of the prior session's contrast level for each subsequent session. Participants will complete 4 x 1-hour sessions per week for two weeks. After 2 weeks of treatment, participants will be offered the opportunity to complete an additional 2 weeks (8 hours) of treatment. Treatment will take place in the home or in-office depending on the study site.

The control group will patch for 2 hours every day, at home, for 2 weeks. A calendar will be provided (to both groups) in order for parents to track compliance. After 2 weeks of patching, participants in the control group have the option to crossover to the treatment group for an additional 2 weeks.

The primary analysis will compare visual acuity improvements from baseline between the binocular treatment and patching groups after 2 weeks of treatment. Secondary analyses will include comparisons of binocular vision and motor function outcomes between the binocular treatment and patching groups, comparisons of at-home vs. in-office binocular treatment outcomes and an evaluation of crossover effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-5.9 years old (36-83 months at the time of registration)
* Confirmed diagnosis of amblyopia
* Best-corrected visual acuity of 20/32 - 20/100 in the amblyopic eye
* Best-corrected visual acuity of 20/16 - 20/40 in fellow eye for ages 3-4, and 20/16-20/32 for ages 5-5.9
* Interocular difference in visual acuity of 3 lines or greater
* If anisometropic, anisometropia (≥1.00D)
* Wearing glasses for 8+ weeks + no change in VA w/ glasses for 4-6 weeks
* Must be able to experience simultaneous perception when viewing the binocular treatment stimuli with an appropriate interocular contrast offset
* Doctor and parent must be willing to forego patching/drops for 4 week study period

Exclusion Criteria:

* strabismus
* Diagnosed eye disease or visual disorder other than amblyopia or anisometropia
* >8 weeks premature
* Diagnosed or suspected developmental delay (eg. learning disability, autism, Down syndrome)
* Diagnosed systemic disease (eg. diabetes, lupus, albinism)

Ages: 36 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 2 weeks
  Change in visual acuity, measured in logMAR using an electronic HOTV test

SECONDARY OUTCOMES:
Visual acuity | 4 weeks
  Change in visual acuity, measured in logMAR an electronic HOTV test
Motor function | 2 weeks
  Change in motor function, measured using the Movement Assessment Battery for Children-2 (version 2)
Stereopsis | 2 weeks
  Change in stereopsis, measured using the Randot Preschool Stereoacuity Test
Treatment adherence | 4 weeks
  Self-reported amount of time spent viewing the cartoon or patching compared to amount of prescribed time
Treatment adherence | 2 weeks
  Self-reported amount of time spent viewing the cartoon or patching compared to amount of prescribed time
Stereopsis | 4 weeks
  Change in stereopsis, measured using the Randot Preschool Stereoacuity Test
Motor function | 4 weeks
  Change in motor function, measured using the Movement Assessment Battery for Children-2 (version 2)
Interocular suppression | 2 weeks
  Change in interocular suppression measured using the Worth 4 dot test
Interocular suppression | 4 weeks
  Change in interocular suppression measured using the Worth 4 dot test
Interocular contrast balance | 2 weeks
  Change in interocular contrast balance measured using a dichoptic letter chart
Interocular contrast balance | 4 weeks
  Change in interocular contrast balance measured using a dichoptic letter chart

CONTACTS AND LOCATIONS:
Overall Officials: Ben Thompson, PhD, Principal Investigator — University of Waterloo
Locations (2):
- Retina Foundation of the Southwest, Dallas, Texas, United States
- Queensland University of Technology, Brisbane, Queesnland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jost RM, Kelly KR, Birch EE. Risk of recurrence after cessation of dichoptic, binocular treatment of amblyopia. J AAPOS. 2023 Oct;27(5):298-300. doi: 10.1016/j.jaapos.2023.06.009. Epub 2023 Aug 23. PMID 37619861